CLINICAL TRIAL: NCT01429155
Title: Post Transplant Course of Hepatitis C Patients After Living Donor Liver Transplant in Association With Interleukin 28 B
Brief Title: Outcomes in Hepatitis C After Living Donor Liver Transplantation in Association With Interleukin 28 B
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Humberto C. Gonzalez, Gastroenterology Fellow, Henry Ford Health System
Other Study IDs: 6975
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C
Keywords: End stage liver disease; Living donor liver transplantation; Hepatitis C; Interleukin 28B
MeSH Terms: conditions — Hepatitis C; End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Liver transplant recipeints: Patients suffering from chronic hepatitis C that required a living donor liver transplant.
  Interventions: Genetic: Interleukin 28B genotype
- Liver Donors: Patients who donated part of their liver to a patient suffering from chronic hepatitis C
  Interventions: Genetic: Interleukin 28B genotype

INTERVENTIONS:
Genetic: Interleukin 28B genotype — Interleukin 28B genotype will be obtained from a tissue block of the liver explant (liver transplanted patients) Interleukin 28B genotype will be obtained from a blood sample drawn (liver donors)

SUMMARY:
Hepatitis C is the leading cause of liver transplants in the USA. Given that there is a national organ shortage, living donor liver transplantation has became a viable option for patients with end stage liver disease who are not severely ill. Recently particular polymorphisms of IL-28B gene were reported to correlate with histological recurrence and antiviral treatment response after orthotopic liver transplantation for hepatitis C. Similar results have not been described yet in living donor liver transplant patients.

There is data suggesting slightly inferior outcomes in living donor liver transplants when done for hepatitis C. The investigators postulate that such inferior outcomes may be related to IL28 polymorphism concordance (i.e., unfavorable recipient polymorphism patients receive similarly unfavorable polymorphism livers from their relatives).

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a living donor liver transplant for chronic hepatitis C who are 18 year or older
* Patients who donated part of their liver to patients suffering from chronic hepatitis C. Donors must be 18 years or older

Exclusion Criteria:

* Patients who are not willing to sign the consent
* Inability to obtain liver specimen (recipients)
* Inability to obtain blood sample (donors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C patients that required a living donor liver transplant will be identified from the liver tranplant registry.
  Living liver donors will be indentified from the liver tranplant registry.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Sustained virological response after living donor liver transplant | 12-24 months
  Determine if sustained virological response is achieved after liver transplantation for hepatitis C with antiviral therapy (rivabirin and pegelated interferon) based on patient IL28B genotype

SECONDARY OUTCOMES:
Liver retransplantation | 1-24 months
  Determine the need of liver retransplantion based on the IL 28B genotype

CONTACTS AND LOCATIONS:
Overall Officials: Humberto C Gonzalez, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Charlton MR, Thompson A, Veldt BJ, Watt K, Tillmann H, Poterucha JJ, Heimbach JK, Goldstein D, McHutchison J. Interleukin-28B polymorphisms are associated with histological recurrence and treatment response following liver transplantation in patients with hepatitis C virus infection. Hepatology. 2011 Jan;53(1):317-24. doi: 10.1002/hep.24074. PMID 21254179
- [Background] Eurich D, Boas-Knoop S, Ruehl M, Schulz M, Carrillo ED, Berg T, Neuhaus R, Neuhaus P, Neumann UP, Bahra M. Relationship between the interleukin-28b gene polymorphism and the histological severity of hepatitis C virus-induced graft inflammation and the response to antiviral therapy after liver transplantation. Liver Transpl. 2011 Mar;17(3):289-98. doi: 10.1002/lt.22235. PMID 21384511